CLINICAL TRIAL: NCT03759951
Title: The Dose-response Effect of High-intensity Interval Neuromuscular Training on Health, Performance and Quality of Life in Overweight/Obese Adults: The DoIT Trial
Brief Title: Hybrid Exercise Training for Health, Performance and Well-Being (DoIT II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DoIT II-UTH
Record Dates: First submitted 2018-11-22; First posted 2018-11-30 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: High-Intensity Interval Training; Body Composition; Performance; Habitual Physical Activity
Keywords: functional training; circuit training; interval training; neuromuscular training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Experimental): No intervention. Participated only in measurements at baseline, at 6 months and at 12 months.
  Interventions: Behavioral: Control
- DoIT-1 (Experimental): Participated in a supervised 1-year workout exercise training program once per week and in measurements at baseline, at 6 months and at 12 months.
  Interventions: Behavioral: DoIT-1
- DoIT-2 (Experimental): Participated in a supervised 1-year workout exercise training program twice per week and in measurements at baseline, at 6 months and at 12 months.
  Interventions: Behavioral: DoIT-2
- DoIT-3 (Experimental): Participated in a supervised 1-year workout exercise training program thrice per week and in measurements at baseline, at 6 months and at 12 months.
  Interventions: Behavioral: DoIT-3

INTERVENTIONS:
Behavioral: DoIT-1 — A hybrid small-group (5-10 participants/session) training modality, that combines interval training, circuit-based resistance exercise and functional training and performed according to a periodized model of exercise prescription as an alternative approach for weight management, health, performance and well-being. DoIT will be performed once per week on non-consecutive days for 12 months.
  Other Names: Hybrid Interval Training
  Arms: DoIT-1
Behavioral: DoIT-2 — A hybrid small-group (5-10 participants/session) training modality, that combines interval training, circuit-based resistance exercise and functional training and performed according to a periodized model of exercise prescription as an alternative approach for weight management, health, performance and well-being. DoIT will be performed twice per week on non-consecutive days for 12 months.
  Other Names: Hybrid Interval Training
  Arms: DoIT-2
Behavioral: DoIT-3 — A hybrid small-group (5-10 participants/session) training modality, that combines interval training, circuit-based resistance exercise and functional training and performed according to a periodized model of exercise prescription as an alternative approach for weight management, health, performance and well-being. DoIT will be performed thrice per week on non-consecutive days for 12 months.
  Other Names: Hybrid Interval Training
  Arms: DoIT-3
Behavioral: Control — No training will be performed during a 1-year period. Participation only in measurements.
  Arms: Control

SUMMARY:
Observing a lack of research investigating the chronic physiological and psychological responses to this type of exercise training the aim of this study is to investigate the optimal training configurations of DoIT to produce positive effects on health, performance and quality of life markers in sedentary overweight or obese adults aged 30-55 years. The DoIT program will be performed in a small-group setting indoor or outdoor implementing a progressive manner for 12 months and using bodyweight exercises with alternative modes.

DETAILED DESCRIPTION:
This controlled, randomized, four-group, repeated-measures clinical trial will be consisted of the following stages:

1. Initial testing: body weight and height, RMR, daily physical activity (PA), daily nutritional intake.
2. a 4-week adaptive period: based on a dietary analysis, participants will be given a dietary plan (considering the RMR and total daily physical activity related energy expenditure), providing an isocaloric diet over the initial 4-week adaptive period. During this adaptive period, volunteers will also be familiarized with exercises techniques and overload patterns that will be used throughout the study through 4 preparatory sessions.
3. At the end of the adaptation period, participants will participate in assessment procedures (baseline testing) at University facilities.
4. After the adaptive period all participants will be randomly assigned to four groups (control, 1 session/week, 2 sessions/week, 3 sessions/week). The exercise protocols that will be used throughout the 1-year intervention will be consisted of 8-12 neuromotor exercises in circuit fashion applying prescribed time (15-45 sec) of effort and passive recovery intervals.
5. After 12 months of exercise intervention all participants will participate in assessment procedures (post-training testing) at University facilities within 5 days after the completion of the last training session.

All participants will be randomly assigned to the following four groups:

1. Control group (no training)
2. DoIT-1 (1 session/week)
3. DoIT-2 (2 sessions/week)
4. DoIT-3 (3 sessions/week)

ELIGIBILITY:
Inclusion Criteria:

1. inactivity (no exercise participation for ≥6 months before the study; VO2max <30 ml·kg-1·min-1)
2. age of 30-55 years
3. overweight/obese (BMI 25.0-39.9)
4. body fat percentage for women > 32% and for men > 25%
5. waist circumference for women > 80 cm and for men > 94 cm
6. medical clearance for strenuous physical training
7. no smoking for ≥6 months before the study
8. no diet intervention or usage of nutritional supplements/medications before (≥6 months) and during the study
9. no weight loss greater >10% of body mass before (≤6 months) the study
10. no diagnosis or symptoms of cardiovascular, metabolic, pulmonary, renal, musculoskeletal or mental disorders

Exclusion Criteria:

Participants will be excluded from the study if they:

1. will not participate in ≥80% of total exercise sessions
2. will adhere to a nutritional intervention during the study
3. will modify the habitual physical activity levels during the study

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in body mass | At baseline, at 6 months and at 12 months
  Body mass (kg) will be measured using a beam scale
Change in body mass index | At baseline, at 6 months and at 12 months
  Body mass index will be calculated using the Quetelet's equation
Change in waist circumference | At baseline, at 6 months and at 12 months
  Waist circumference (cm) will be measured using a Gullick II tape
Change in hip circumference | At baseline, at 6 months and at 12 months
  Hip circumference (cm) will be measured using a Gullick II tape
Change in waist-to-hip ratio | At baseline, at 6 months and at 12 months
  Waist-to-hip ratio will be calculated by dividing the waist by the hip measurement
Change in body fat | At baseline and at 12 months
  Body fat (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Change in fat mass | At baseline and at 12 months
  Body fat (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Change in fat-free mass | At baseline and at 12 months
  Fat-free mass (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Change in resting metabolic rate (RMR) | At baseline, at 6 months and at 12 months
  RMR (kcal) will be measured using a portable open-circuit indirect calorimeter with a ventilated hood system
Change in maximal strength (1RM) | At baseline, at 6 months and at 12 months
  1RM (kg) for the lower body will be measured bilaterally on a horizontal leg press, seated leg extension and lying leg curl machines while 1RM (kg) for the upper body will be measured on a seated chest press and lat pull-down machines
Change in maximal oxygen consumption (VO2max) | At baseline, at 6 months and at 12 months
  VO2max (ml/kg/min) will be estimated using a low-risk, low-cost and single-stage submaximal treadmill walking test
Change in habitual physical activity (PA) | At baseline, at 3, 6, 9 and 12 months
  Seven-day habitual PA (MET-min/week) will be assessed using the International Physical Activity Questionnaire (IPAQ)
Change in dietary intake | At baseline, at 3, 6, 9 and 12 months
  Dietary intake (kcal) will be assessed using 7-day diet recalls
Change in body mass content (BMC) | At baseline and at 12 months
  BMC (g) will be assessed by dual-energy X-ray absorptiometry (DXA) of the total body and non-dominant hip.
Change in body mass density (BMD) | At baseline and at 12 months
  BMD (g) will be assessed by dual-energy X-ray absorptiometry (DXA) of the total body and non-dominant hip.
Change in resting systolic (SBP) and diastolic (DBP) blood pressures. | At baseline, at 6 months and at 12 months
  Resting SBP (mmHg) and DBP (mmHg) will be assessed by a manual sphygmomanometer
Change in mean arterial pressure (MAP). | At baseline, at 6 months and at 12 months
  MAP (mmHg) will be calculated using the following equation: MAP = SBP + (DBP × DBP) / 3
Change in resting heart rate (RHR). | At baseline, at 6 months and at 12 months
  RHR (bpm) will be measured by pulse palpation for 60 seconds.
Change in muscular endurance | At baseline, at 6 months and at 12 months
  Muscular endurance (repetitions until muscle failure) will be assessed using timed tests (60 sec) for the abdominal musculature, upper and lower body. The tests will include partial curl-up, push-up for males and modified push-up for females (kneeling position) and modified chair squat, respectively
Change in flexibility | At baseline, at 6 months and at 12 months
  Flexibility (cm) will be assessed using the modified sit-and-reach test
Change in static balance | At baseline, at 6 months and at 12 months
  Static balance (sec) will be assessed using the Sharpened Romberg test
Change in functional capacity | At baseline, at 6 months and at 12 months
  Functional capacity will be assessed using a movement-based screening tool titled Functional Movement Screening (FMS). The FMS will be consisted of 7 movement tasks that will be scored from 0 to 3 points and the sum will create score ranging from 0 to 21 points (0 = pain with pattern regardless of quality, 1 = unable to perform pattern, 2 = able to perform pattern with compensation/imperfection, 3 = able to perform pattern as directed).
Change in blood lipids | At baseline and at 12 months
  Total serum cholesterol (mmol/L), triglycerides (mmol/L), low-density lipoprotein (mmol/L) and high-density lipoprotein (mmol/L) will be measured with commercially availlable kits
Change in blood inflammatory markers | At baseline and at 12 months
  Cytokines, lipocalines, CRP, oxidative stress markers will be measured with commercially availlable kits
Change in cortisol | At baseline and at 12 months
  Cortisol (nmol/L) will be measured with commercially availlable kits
Change in insulin | At baseline and at 12 months
  Insulin (mIU/L) will be measured with commercially availlable kits
Change in homeostatic model assessment for insulin resistance (HOMA-IR) | At baseline and at 12 months
  HOMA-IR will be measured with commercially availlable kits. ΗΟΜΑ score will be calculated using the equation HOMA-IR = fasting insulin (mIU/L) x fasting glucose (mg/dL) / 405. HOMA-IR score will be classified using the following range: normal insulin resistance < 3, moderate insulin resistance 3-5, severe insulin resistance > 5)
Change in leptin | At baseline and at 12 months
  Leptin (μg/L) will be measured with commercially availlable kits
Change in adiponectin | At baseline and at 12 months
  Adiponectin (μg/mL) will be measured with commercially availlable kits
Change in interleukin 1 beta (IL-1b) and interleuking 6 (IL-6) | At baseline and at 12 months
  IL-1b and IL-6 (pg/ml) will be measured with commercially availlable kits
Change in fasting blood glucose (FBG) | At baseline and at 12 months
  FBG (mg/dL) will be measured with commercially availlable kits
Change in serum protein carbonyl levels | At baseline and at 12 months
  Protein carbonyl (mg) will be measured with commercially availlable kits
Change in thiobarbituric acid-reactive substances (TBARS) | At baseline and at 12 months
  TBARS (nmol/mg protein) will be measured with commercially availlable kits
Change in reduced (GSH) and oxidized (GSSG) glutathione | At baseline and at 12 months
  GSH and GSSG (nmol/L) will be measured with commercially availlable kits
Change in catalase activity | At baseline and at 12 months
  Catalase activity (units) will be measured with commercially availlable kits
Change in total antioxidant capacity (TAC) | At baseline and at 12 months
  TAC (mmol/l) will be measured with commercially availlable kits
Change in C-reactive protein (CRP) | At baseline and at 12 months
  CRP (mg/L) will be measured with commercially availlable kits
Change in cholecystokinin (CKK) | At baseline and at 12 months
  CKK (ng/ml) will be measured with commercially availlable kits
Change in pancreatic polypeptide (PP) | At baseline and at 12 months
  PP (pg/ml) will be measured with commercially availlable kits
Change in peptide YY (PYY) | At baseline and at 12 months
  PYY (ng/ml) will be measured with commercially availlable kits
Change in oxyntomodulin (OXM) | At baseline and at 12 months
  OXM (pg/ml) will be measured with commercially availlable kits
Change in ghrelin | At baseline and at 12 months
  Ghrelin (pg/ml) will be measured with commercially availlable kits
Change in glucagon-like peptide-1 (GLP-1) | At baseline and at 12 months
  GLP-1 (pg/ml) will be measured with commercially availlable kits
Change in appetite | At baseline, at 6 months and at 12 months
  The Visual Analog Scale (VAS) will be used to measure perceived hunger, satiety, and individual's own interpretation of their hunger sensations. VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured orientated from the left (worst) to the right (best).
Change in quality of life | At baseline, at 6 months and at 12 months
  Quality of life will be assessed using the physical and mental component subscales of the Greek 36-Item Short-Form Health Survey (SF-36). The scores on both component subscales of the SF-36 will range from 0 to 100, with higher scores indicating better health status while the minimal clinically important difference will be 2 points.
Change in exercise enjoyment | At baseline, at 6 months and at 12 months
  Exercise enjoyment will be assessed using the Exercise Enjoyment Scale (EES), which is a single-item 7-point scale to assess enjoyment pre-, during, and post-exercise ranging from "not at all" at 1 to "extremely" at 7.
Change in affective valence | At baseline, at 6 months and at 12 months
  Affective responses to exercise will be assessed using the Feeling Scale (FS), which is a single-item 11-point scale to assess feeling of pleasure pre-, during, and post-exercise training ranging from "very good" at -5 to "very bad" at 5.
Change in irisin | At baseline and at 12 months
  Irisin (ng/ml) will be measured with commercially availlable kits
Change in left ventricular end-diastolic volume (LVEDV). | At baseline and at 12 months
  LVEDV (ml) will be measured using echocardiography.
Change in left ventricular end-systolic volume (LVESV). | At baseline and at 12 months
  LVESV (ml) will be measured using echocardiography.
Change in left ventricular stroke volume (LVSV). | At baseline and at 12 months
  LVSV (ml) will be measured using echocardiography.
Change in interventricular septum end diastole (IVSd). | At baseline and at 12 months
  IVSd (mm) will be measured using echocardiography.
Change in interventricular septum end diastole (IVSs). | At baseline and at 12 months
  IVSs (mm) will be measured using echocardiography.
Change in left ventricular ejection fraction (LVEF). | At baseline and at 12 months
  LVEF (%) will be measured using echocardiography.
Change in left ventricular internal diameter end diastole (LVIDd). | At baseline and at 12 months
  LVIDd (mm) will be measured using echocardiography.
Change in left ventricular internal diameter end systole (LVIDs). | At baseline and at 12 months
  LVIDs (mm) will be measured using echocardiography.
Change in left ventricular posterior wall end diastole (LVPWd). | At baseline and at 12 months
  LVPWd (mm) will be measured using echocardiography.
Change in left ventricular mass (LV mass). | At baseline and at 12 months
  LV mass (g) will be measured using echocardiography.
Change in left atrial (LA) diameter. | At baseline and at 12 months
  LA diameter (mm) will be measured using echocardiography.
Change in aortic root. | At baseline and at 12 months
  Aortic root (mm) will be measured using echocardiography.
Change in aortic valve velocity (AoV Vel). | At baseline and at 12 months
  AoV Vel (cm/s) will be measured using echocardiography.
Change in aortic valve pressure gradient (AoV PG). | At baseline and at 12 months
  AoV PG (mmHg) will be measured using echocardiography.
Change in right ventricular end diastole (RVD). | At baseline and at 12 months
  RVD (mm) will be measured using echocardiography.
Change in pulmonary artery systolic pressure (PASP). | At baseline and at 12 months
  PASP (mmHg) will be measured using echocardiography.
Change in left ventricular fractional shortening (FS). | At baseline and at 12 months
  Fractional shortening (%) will be measured using echocardiography.
Change in depression II. | At baseline, at 6 months and at 12 months
  Depression will be measured using the Patient Health Questionnaire (PHQ-9)), which is a self-administered instrument consisiting of 9 multiple-choice questions scored from 0 to 3. Higher total scores indicate higher depression severity.
Change in depression I. | At baseline, at 6 months and at 12 months
  Depression will be measured using the Beck Depression Inventory (BDI), which is a self-report questionnaire consisiting of 21 multiple-choice questions scored from 0 to 3. Higher total scores indicate more severe depressive symptoms.
Change in depression and anxiety. | At baseline, at 6 months and at 12 months
  Both depression and anxiety will be measured using the Hospital Anxiety and Depression Scale (HADS), which is a 14-item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Higher scores indicate greater anxiety and depression.
Change in mood. | At baseline, at 6 months and at 12 months
  Mood will be measured using the Profile of Mood States (POMS) questionnaire, which uses a unipolar scale to rate the extent to which they are experiencing or have experienced 20 affect states in the past week using a 5-point scale (0 = not at all, 4 = extremely). Higher scores indicate greater negative mood.
Change in anxiety. | At baseline, at 6 months and at 12 months
  Anxiety will be measured using the State-Trait Anxiety Inventory (STAI), which is an instrument that has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Change in physical self. | At baseline, at 6 months and at 12 months
  Physical self will be measured using the Physical Self-Perception Profile (PSPP), which is an instrument with 30 questions comprising five 6-item subscales. Each item has a four-point structured-alternative format. Scores range from 6 to 24 on each subscale, with high scores representing positive perceptions. Half of the items are worded in the negative direction.

SECONDARY OUTCOMES:
Change in exercise-induced caloric expenditure | At baseline, at 6 months and at 12 months
  Measured using a portable indirect calorimetry system
Change in blood lactate concentration (BLa) | At baseline, at 6 months and at 12 months
  BLa (mmol/L) concentration will be measured in a microphotometer with commercially available kits. Blood samples will be collected pre-, mid- and post-exercise session (single bout) at 3 min post-exercise
Change in peak expiratory flow (PEF) | At baseline and at 12 months
  PEF (l/s) will be measured using the maximum flow volume loop.
Change in forced expiratory flow between 25 and 75% of vital capacity (FEF25-75). | At baseline and at 12 months
  FEF25-75 (l/s) will be measured using the maximum flow volume loop.
Change in forced expiratory volume at 1 s (FEV1). | At baseline and at 12 months
  FEV1 (l) will be measured using the maximum flow volume loop.
Change in forced vital capacity (FVC). | At baseline and at 12 months
  FVC (l) will be measured using the maximum flow volume loop.
Change in the ratio of FEV1/FVC. | At baseline and at 12 months
  FEV1/FVC (%) will be measured using the maximum flow volume loop.

CONTACTS AND LOCATIONS:
Overall Officials: Alexios Batrakoulis, MSc, Principal Investigator — SmArT Lab, DPESS, University of Thessaly
Locations (1):
- Laboratory of Exercise Physiology, Exercise Biochemistry and Sports Nutrition, School of Physical Education, Sports Sciences and Dietetics, University of Thessaly, Trikala, Greece

REFERENCES:
- [Background] Batrakoulis A, Fatouros IG, Chatzinikolaou A, Draganidis D, Georgakouli K, Papanikolaou K, Deli CK, Tsimeas P, Avloniti A, Syrou N, Jamurtas AZ. Dose-response effects of high-intensity interval neuromuscular exercise training on weight loss, performance, health and quality of life in inactive obese adults: Study rationale, design and methods of the DoIT trial. Contemp Clin Trials Commun. 2019 May 23;15:100386. doi: 10.1016/j.conctc.2019.100386. eCollection 2019 Sep. PMID 31193901
- [Result] Batrakoulis A, Jamurtas AZ, Tsimeas P, Poulios A, Perivoliotis K, Syrou N, Papanikolaou K, Draganidis D, Deli CK, Metsios GS, Angelopoulos TJ, Feito Y, Fatouros IG. Hybrid-type, multicomponent interval training upregulates musculoskeletal fitness of adults with overweight and obesity in a volume-dependent manner: A 1-year dose-response randomised controlled trial. Eur J Sport Sci. 2023 Mar;23(3):432-443. doi: 10.1080/17461391.2021.2025434. Epub 2022 Jan 31. PMID 34974824